CLINICAL TRIAL: NCT06838104
Title: Effect of Melatonin on Positive and Negative Symptoms of Schizophrenic Patients: a Randomized Placebo-Controlled Study
Brief Title: Effect of Melatonin on Schizophrenic Symptoms: a Randomized Placebo-Controlled Trial
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lahore General Hospital (Other Government)
Responsible Party: Principal Investigator, Muhammad Irfan Jamil, Principal Investigator, Lahore General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LahoreGeneralH2
Record Dates: First submitted 2025-02-15; First posted 2025-02-20 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Schizophrenia Disorders; Psychotic Disorder
Keywords: Antipsychotic Therapy; Positive Symptoms; Negative Symptoms
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Melatonin (Experimental): will receive 6 mg of melatonin orally, administered as two 3 mg tablets 30 minutes before bedtime daily for 8 weeks, alongside their standard antipsychotic treatment (risperidone 6-8 mg/day).
  Interventions: Drug: Melatonin
- Placebo (Placebo Comparator): will receive placebo tablets identical in shape, size, smell, taste, and color to melatonin tablets, administered in the same manner (two tablets 30 minutes before bedtime) for 8 weeks, alongside their standard antipsychotic treatment (risperidone 6-8 mg/day).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Melatonin — Participants in this group will receive 6 mg of melatonin orally, administered as two 3 mg tablets 30 minutes before bedtime daily for 8 weeks, alongside their standard antipsychotic treatment (risperidone 6-8 mg/day).
  Arms: Melatonin
Drug: Placebo — Participants in this group will receive placebo tablets identical in shape, size, smell, taste, and color to melatonin tablets, administered in the same manner (two tablets 30 minutes before bedtime) for 8 weeks, alongside their standard antipsychotic treatment (risperidone 6-8 mg/day).
  Arms: Placebo

SUMMARY:
Schizophrenia is a chronic mental health disorder that affects thoughts, emotions, and behaviors. It includes positive symptoms such as hallucinations and delusions, as well as negative symptoms like reduced motivation, social withdrawal, and blunted emotional expression.

This study is a randomized, placebo-controlled trial designed to evaluate the effect of melatonin on schizophrenia symptoms. Melatonin, a natural hormone that regulates sleep, has antioxidant properties and potential neuroprotective effects.

A total of 76 patients diagnosed with schizophrenia according to DSM-5 criteria will be randomly assigned to receive either melatonin (6 mg daily) or a placebo for eight weeks while continuing their standard risperidone-based antipsychotic therapy. Symptoms will be assessed at baseline and after 8 weeks using the Positive and Negative Syndrome Scale (PANSS), a validated tool for measuring schizophrenia severity. The primary outcome will be changes in PANSS scores, evaluating whether melatonin leads to significant improvement compared to placebo.

The study hypothesizes that melatonin will significantly reduce positive and negative symptoms compared to placebo. Findings from this research may help determine whether melatonin can be used as an adjunctive treatment in schizophrenia, potentially improving clinical outcomes and quality of life for patients.

DETAILED DESCRIPTION:
Schizophrenia is a chronic psychiatric disorder characterized by a combination of positive symptoms (hallucinations, delusions, disorganized thinking) and negative symptoms (social withdrawal, reduced motivation, and blunted affect). While antipsychotic medications remain the primary treatment, they often fail to address negative symptoms, which are strongly associated with poor functional prognosis and reduced quality of life. Emerging evidence suggests that melatonin, a neurohormone primarily responsible for sleep regulation, possesses antioxidant and neuroprotective properties that may contribute to symptom improvement in schizophrenia.

This randomized, placebo-controlled trial aims to evaluate the efficacy of melatonin supplementation as an adjunct to standard antipsychotic therapy (risperidone 6-8 mg/day) in patients diagnosed with schizophrenia. The study will enroll 76 patients, randomly assigned to receive either melatonin (6 mg daily, administered as two 3 mg tablets before bedtime) or a placebo identical in shape, size, color, and taste for eight weeks. Participants will continue their standard antipsychotic regimen throughout the study period.

The primary outcome of the study is the change in Positive and Negative Syndrome Scale (PANSS) total score from baseline to week 8, assessing the overall impact of melatonin on symptom severity. The secondary outcomes include changes in PANSS negative symptom subscale scores, evaluating whether melatonin improves motivation, emotional expression, and social engagement.

To ensure methodological rigor, patients will be assessed at baseline and after eight weeks using the PANSS scoring system. Randomization will be performed using a lottery method, and the study will follow a double-blind design, ensuring that neither patients nor investigators are aware of the treatment allocation. Safety monitoring will include adverse event reporting, particularly evaluating the incidence of excessive sedation, dizziness, headache, and gastrointestinal disturbances.

This study aims to provide clinical evidence regarding the role of melatonin as an adjunctive treatment for schizophrenia. If proven effective, melatonin supplementation could offer a low-cost, well-tolerated intervention to enhance treatment outcomes in schizophrenia patients, particularly those experiencing persistent negative symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 to 50 years.
* Patients diagnosed with schizophrenia according to DSM-5 criteria, exhibiting both positive negative symptoms.
* Patients who score less than 6 on the Calgary Depression Scale for Schizophrenia (CDSS), indicating no significant depressive episode, will be considered eligible.

Exclusion Criteria:

* Patients with a known hypersensitivity or allergy to melatonin or any of its excipients.
* Patients with a current or past diagnosis of major depressive disorder, bipolar disorder, or obsessive-compulsive disorder, unless these are in full remission and do not require active pharmacological treatment.
* Patients with any unstable or serious medical condition (e.g., cardiovascular, hepatic, renal, or respiratory diseases) that could interfere with the study outcomes or pose additional risk to the patient.
* Married women of reproductive age, unless they use a reliable non-hormonal contraception method.
* Patients with neurological disorders, such as epilepsy, Parkinson's disease, or traumatic brain injury, which may mimic psychiatric symptoms.
* Use of antiepileptic, antihypertensive, anticoagulant, or anti-platelet drugs.
* Use of inhibitors or stimulants of hepatic isoenzymes that metabolize melatonin or olanzapine (e.g., omeprazole, rifampin, fluvoxamine, ciprofloxacin, carbamazepine, modafinil).
* History of addictive disorders.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2024-12-05 (Actual); Primary Completion 2025-06-05 (Estimated); Study Completion 2025-06-05 (Estimated)

PRIMARY OUTCOMES:
Change in Positive and Negative Syndrome Scale (PANSS) Total Score | Baseline (Week 0) and Week 8
  The PANSS is a standardized tool used to measure the severity of schizophrenia symptoms, including positive symptoms (hallucinations, delusions), negative symptoms (social withdrawal, lack of motivation), and general psychopathology symptoms. The primary outcome will be the mean change in PANSS total score from baseline to the 8-week follow-up, assessing the effectiveness of melatonin in reducing schizophrenia symptoms.

SECONDARY OUTCOMES:
Change in PANSS Negative Symptom Subscale Score | Baseline (Week 0) and Week 8
  The PANSS negative symptom subscale consists of seven items, measuring deficits in emotional expression, motivation, speech, and social engagement. The score ranges from 7 to 49, with higher scores reflecting more severe negative symptoms. The mean change from baseline to Week 8 will be analyzed to assess the impact of melatonin on negative symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Irfan Jamil, Principal Investigator — Lahore General Hospital, Lahore
Locations (1):
- Lahore General Hospital, Lahore, Lahore, Punjab Province, Pakistan